CLINICAL TRIAL: NCT07140146
Title: Comparison of Trehalose and Glycine Air-Polishing Powders in the Supportive Treatment of Peri-Implant Mucositis and Their Effect on Implant Surface Integrity: A Randomized Controlled Clinical Trial
Brief Title: Trehalose vs Glycine Air-Polishing in Peri-Implant Mucositis Treatment
Acronym: TREAL-G
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-TREALOSEIMPLANT
Record Dates: First submitted 2025-07-19; First posted 2025-08-24 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Peri-implant Mucositis
Keywords: Peri-Implant Mucositis; Trehalose Powder; Glycine Powder; Air Polishing; Dental Implants; Implant Surface Integrity; Biofilm Removal; Randomized Controlled Trial; Scanning Electron Microscopy (SEM)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trehalose Powder Air-Polishing with Supportive Peri-Implant Therapy (Experimental): Patients receive supragingival and subgingival air-polishing with trehalose powder in combination with supportive peri-implant therapy, including manual and ultrasonic debridement, at baseline, 1, 3, and 6 months. Clinical parameters evaluated include Plaque Index (PI), Bleeding on Probing (BoP), Probing Pocket Depth (PPD), and Bleeding Score (BS). In vitro scanning electron microscopy (SEM) is used to assess potential alterations on the implant surface.
  Interventions: Device: Trehalose Powder Air-Polishing
- Glycine Powder Air-Polishing with Supportive Peri-Implant Therapy (Active Comparator): Patients receive supragingival and subgingival air-polishing with glycine powder in combination with supportive peri-implant therapy, including manual and ultrasonic debridement, at the same timepoints (baseline, 1, 3, and 6 months). The same clinical parameters (PI, BoP, PPD, BS) are recorded. Implant surface integrity is assessed post-treatment by scanning electron microscopy (SEM).
  Interventions: Device: Glycine Powder Air-Polishing

INTERVENTIONS:
Device: Trehalose Powder Air-Polishing — Air-polishing procedure using trehalose-based powder (particle size <65 µm, low abrasiveness) applied supra- and subgingivally with a professional air-polishing device in patients diagnosed with peri-implant mucositis. The intervention is combined with non-surgical debridement using manual curettes and ultrasonic scalers. The procedure is performed at baseline (T0), and repeated at 1 month (T1), 3 months (T2), and 6 months (T3). Clinical outcomes assessed include Plaque Index (PI), Bleeding on Probing (BoP), Probing Pocket Depth (PPD), and Bleeding Score (BS). Implant surfaces are also evaluated in vitro using scanning electron microscopy (SEM) to assess any surface alterations after powder application.
  Arms: Trehalose Powder Air-Polishing with Supportive Peri-Implant Therapy
Device: Glycine Powder Air-Polishing — Air-polishing procedure using glycine-based powder (particle size ~25 µm, amino acid composition) applied supra- and subgingivally with a professional air-polishing device in patients with peri-implant mucositis. This treatment is combined with standard non-surgical supportive peri-implant therapy involving manual and ultrasonic debridement. The procedure is performed at baseline (T0), and repeated at 1 month (T1), 3 months (T2), and 6 months (T3). The intervention aims to reduce plaque accumulation and inflammation. Clinical parameters recorded include PI, BoP, PPD, and BS. Implant surfaces are also assessed in vitro via SEM to compare the effects of glycine versus trehalose on implant surface integrity.
  Arms: Glycine Powder Air-Polishing with Supportive Peri-Implant Therapy

SUMMARY:
This randomized controlled clinical trial investigates the effectiveness of trehalose powder compared to glycine powder when used in air-polishing during supportive therapy for peri-implant mucositis, a reversible inflammatory condition affecting the soft tissues around dental implants.

A total of 40 adult patients with peri-implant mucositis will be enrolled and randomly assigned to receive non-surgical periodontal therapy combined with air-polishing using either trehalose powder (test group) or glycine powder (control group). Clinical parameters will be evaluated at baseline, 1 month, 3 months, and 6 months. These include Plaque Index (PI), Bleeding on Probing (BoP), Probing Pocket Depth (PPD), and Bleeding Score (BS), in order to assess plaque accumulation, inflammation, and bleeding.

The primary objective is to compare the reduction in plaque levels between the two groups over the study period. Secondary outcomes include evaluation of changes in gingival inflammation and probing depths, as well as assessment of implant surface integrity through in vitro scanning electron microscopy (SEM) after treatment.

The aim of the study is to determine whether trehalose powder offers improved clinical outcomes and greater implant surface preservation compared to glycine powder in the non-surgical management of peri-implant mucositis.

DETAILED DESCRIPTION:
Peri-implant mucositis is a reversible inflammatory condition affecting the soft tissues surrounding dental implants and represents an early stage in the progression toward peri-implantitis if left untreated. Mechanical debridement combined with minimally invasive biofilm removal strategies has become the cornerstone of current supportive therapy. Among the available options, air-polishing powders have shown favorable outcomes in biofilm disruption without damaging implant surfaces or peri-implant tissues.

This randomized controlled clinical trial aims to compare the clinical efficacy and safety of trehalose powder versus glycine powder in supportive treatment of peri-implant mucositis. Trehalose is a disaccharide with documented antioxidant, anti-inflammatory, and cytoprotective properties, potentially enhancing tissue healing. Glycine, an amino acid widely used in air-polishing, has proven effective in biofilm removal with high biocompatibility and minimal abrasiveness.

Forty patients diagnosed with peri-implant mucositis will be randomly assigned to two groups: a test group receiving supportive periodontal therapy plus air-polishing with trehalose powder, and a control group receiving the same protocol with glycine powder. Clinical outcomes, including plaque accumulation, bleeding on probing, probing pocket depth, and bleeding score, will be assessed at baseline and at 1, 3, and 6 months. In addition, in vitro scanning electron microscopy (SEM) will evaluate implant surface integrity after treatment.

The study is designed to provide new clinical and morphological evidence on the potential benefits of trehalose in peri-implant maintenance protocols and to clarify whether it may represent a valid alternative to glycine for long-term implant health.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 70 years
* Presence of peri-implant mucositis, defined as bleeding on probing (BoP) around implants without radiographic evidence of bone loss beyond initial remodeling
* Visible biofilm on implant surfaces
* Ability to understand and sign informed consent
* Good oral hygiene and patient compliance
* Availability for all follow-up visits (1, 3, and 6 months)

Exclusion Criteria:

* Presence of systemic conditions that may affect healing (e.g., uncontrolled diabetes, immunosuppression)
* Current smokers or former smokers who quit less than 6 months ago
* Pregnant or breastfeeding women
* Use of antibiotics or anti-inflammatory drugs in the 3 months prior to baseline
* Presence of peri-implantitis (i.e., bleeding on probing with concomitant radiographic bone loss)
* History of head and neck radiotherapy
* Presence of pacemakers or cardiac stimulators
* Neurological or psychological disorders affecting study compliance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-30 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Change in plaque accumulation assessed by Plaque Index (PI) | Baseline (T0), 1 month (T1), 3 months (T2), and 6 months (T3)
  The Plaque Index (PI) will be used to assess the amount of bacterial plaque on peri-implant surfaces in patients with peri-implant mucositis. The PI will be recorded on four surfaces per implant (mesial, distal, buccal, and palatal/lingual) following application of a plaque disclosing agent. Scores will be assigned according to a standardized ordinal scale: score 0 indicates no plaque; score 1 corresponds to a thin film of plaque detectable only with a disclosing agent or upon probing; score 2 indicates a moderate accumulation of soft deposits visible to the naked eye; and score 3 reflects abundant plaque deposits on the gingival margin and adjacent implant surfaces. The PI for each implant will be calculated as the mean of the four site-specific scores. The primary endpoint is the difference in mean PI scores between the trehalose and glycine groups across all timepoints. Outcome assessors will be calibrated and blinded to group allocation.

SECONDARY OUTCOMES:
Change in peri-implant inflammation assessed by Bleeding on Probing (BoP) | Baseline (T0), 1 month (T1), 3 months (T2), and 6 months (T3)
  Bleeding on Probing (BoP) will be used to assess peri-implant soft tissue inflammation in patients with peri-implant mucositis. BoP will be recorded by gently probing six sites per implant (mesio-buccal, mid-buccal, disto-buccal, mesio-palatal/lingual, mid-palatal/lingual, disto-palatal/lingual) using a standardized periodontal probe. A positive BoP score is assigned if bleeding occurs within 30 seconds after probing. Each site is scored as either 0 (no bleeding) or 1 (bleeding present). The BoP percentage per implant is calculated as the number of bleeding sites divided by the total number of sites examined (×100). The outcome measure will compare the mean BoP percentages between the Trehalose and Glycine groups across all timepoints. Clinical assessments will be performed by calibrated and blinded investigators.
Change in peri-implant probing depth assessed by Probing Pocket Depth (PPD) | Baseline (T0), 1 month (T1), 3 months (T2), and 6 months (T3)
  Probing Pocket Depth (PPD) will be used to evaluate changes in peri-implant sulcus depth, an indicator of soft tissue inflammation and healing. PPD will be measured using a standardized millimeter-graded periodontal probe at six sites per implant: mesio-buccal, mid-buccal, disto-buccal, mesio-palatal/lingual, mid-palatal/lingual, and disto-palatal/lingual. The probe is inserted parallel to the long axis of the implant, and the distance from the gingival margin to the base of the sulcus is recorded in millimeters. The mean PPD per implant will be calculated and compared between the Trehalose and Glycine groups at all study timepoints. Measurements will be performed by calibrated and blinded examiners.
Change in gingival bleeding severity assessed by Bleeding Score (BS) | Baseline (T0), 1 month (T1), 3 months (T2), and 6 months (T3)
  The Bleeding Score (BS) quantifies the severity of bleeding upon probing in peri-implant tissues. It will be recorded at each implant site showing a positive BoP response, based on the following scale: score 1 indicates minimal bleeding (isolated point), score 2 indicates moderate bleeding (line or triangle of blood), and score 3 indicates profuse bleeding (immediate blood flow covering the implant surface). The BS per implant is calculated as the mean of all site-specific scores. The outcome compares mean BS values between the Trehalose and Glycine groups at each timepoint. All probing will be performed by calibrated, blinded clinicians using gentle pressure.
Changes in implant surface morphology assessed by Scanning Electron Microscopy (SEM) | 6 months (T3)
  Scanning Electron Microscopy (SEM) will be used to evaluate potential morphological changes on implant surfaces after treatment with trehalose or glycine powder. In vitro tests will be conducted using standard titanium dental implant fixtures treated separately with either trehalose or glycine powder under identical air-polishing protocols. After treatment, implants will be cleaned, fixed, and analyzed using a high-resolution desktop SEM system. Surface alterations such as scratches, loss of microstructure, or contaminant residues will be assessed qualitatively and compared descriptively between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, Associate Professor, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the corresponding authors.